CLINICAL TRIAL: NCT04108910
Title: Reduction in Morbidity Rate for Urinary Tract Infections Through Use of PCR-Based Diagnosis and Management
Brief Title: Morbidity Rate for UTI Through Use of PCR-Based Diagnosis and Management
Status: Completed | Type: Observational
Sponsor: Pathnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019 R-VPA-HUS
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Urinary Tract Infections
Keywords: UTI; Home Care
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traditional Urine Culture: Patients treated based upon traditional urine culture
- Guidance PCR/Pooled Sensitivity: Patients treated based upon multiplex UTI PCR/pooled sensitivity results
  Interventions: Diagnostic Test: Guidance UTI

INTERVENTIONS:
Diagnostic Test: Guidance UTI
  Groups: Guidance PCR/Pooled Sensitivity

SUMMARY:
This retrospective study is to determine if the use of PCR for detection and identification of pathogens in UTI along with antimicrobial susceptibility information, affords more efficacious treatment of UTI, as compared to traditional urine culture for patients served by House Call Physicians.

DETAILED DESCRIPTION:
The objective of this study is to determine if retrospective data will show that use of PCR for detection and identification of pathogens in UTI, and antimicrobial susceptibility information, affords more efficacious treatment of UTI, thereby reducing UTI-related morbidity and costs in a patient population that is served by House Call Physicians. House call physicians attend elderly and other adults patients who are suffering from illness or chronic conditions in the safety, privacy, and comfort of their home or assisted living location. In making house calls, physicians ease the burden and difficulty of these chronic patients from traveling to the doctor's office.

ELIGIBILITY:
Inclusion Criteria:

* All patients that the House Call Physician suspects the patient has a UTI and are tagged with the following codes within the medical record

Exclusion Criteria:

* Records where the NPI does not match a known provider or the office listed is not a Specific Population
* Hospice patients
* Records for which DX codes of "X" and "NoDx" where there isn't a diagnostic description.

Ages: 18 Years to 111 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are visited by a House Call Physician and attend to elderly and other adults patients who are suffering from illness or chronic conditions in the safety, privacy, and comfort of their home or assisted living location.
Sampling Method: Non-Probability Sample
Enrollment: 66381 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
ER Visits and or Hospital Admission Rate within 30 days of initial visit related to UTI | 18 Months
  Examine retrospective data of a House Call Patient population to determine if use of PCR, compared with conventional urine culture, leads to a reduction in UTI-related morbidity, as measured by the composite variable number of emergency room/urgent care clinic visits plus the number of admissions to hospital within 30 days of an initial presentation for UTI.

SECONDARY OUTCOMES:
Examine retrospective data to determine if use of PCR, compared with conventional urine culture, leads to a reduction in UTI-related morbidity. | 18 Months
  Examine retrospective data to determine if use of PCR, compared with conventional urine culture, leads to a reduction in UTI-related morbidity:
  * As measured by the number of emergency room visits within 30 days of an initial presentation for UTI.
  * As measured by the number of urgent care clinic visits within 30 days of an initial presentation for UTI.
  * As measured by the number of cases escalated from an urgent care clinic to an emergency room within 30 days of an initial presentation for UTI.
  * As measured by the number of admissions to hospital within 30 days of initial presentation for UTI.
  * As measured by the total hospital length of stay resulting from hospital admission within 30 days of initial presentation for UTI.

OTHER OUTCOMES:
Identify the frequency of observed polymicrobial infections | 18 Months
  Identify the frequency of observed polymicrobial infections (defined as two or more simultaneous bacterial infections), as determined by PCR testing, will be estimated for the population of patients with panel-confirmed UTIs.
  Identify and compare the range and frequency of bacteria species detected by PCR or Traditional Culture within the population of patients.
  Determine if use of PCR and pooled sensitivity provides a different number of options for antibiotic treatment.
  Determine if specific bacteria are more commonly associated with hospital admissions.
  Determine if specific bacteria are more commonly associated with longer length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Wojno, MD, Principal Investigator — Visiting Physicians Association

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suskind AM, Saigal CS, Hanley JM, Lai J, Setodji CM, Clemens JQ; Urologic Diseases of America Project. Incidence and Management of Uncomplicated Recurrent Urinary Tract Infections in a National Sample of Women in the United States. Urology. 2016 Apr;90:50-5. doi: 10.1016/j.urology.2015.11.051. Epub 2016 Jan 26. PMID 26825489
- [Background] Simmering JE, Tang F, Cavanaugh JE, Polgreen LA, Polgreen PM. The Increase in Hospitalizations for Urinary Tract Infections and the Associated Costs in the United States, 1998-2011. Open Forum Infect Dis. 2017 Feb 24;4(1):ofw281. doi: 10.1093/ofid/ofw281. eCollection 2017 Winter. PMID 28480273
- [Background] Qiang XH, Yu TO, Li YN, Zhou LX. Prognosis Risk of Urosepsis in Critical Care Medicine: A Prospective Observational Study. Biomed Res Int. 2016;2016:9028924. doi: 10.1155/2016/9028924. Epub 2016 Feb 3. PMID 26955639
- [Background] Gharbi M, Drysdale JH, Lishman H, Goudie R, Molokhia M, Johnson AP, Holmes AH, Aylin P. Antibiotic management of urinary tract infection in elderly patients in primary care and its association with bloodstream infections and all cause mortality: population based cohort study. BMJ. 2019 Feb 27;364:l525. doi: 10.1136/bmj.l525. PMID 30814048
- [Background] Hsiao CY, Yang HY, Chang CH, Lin HL, Wu CY, Hsiao MC, Hung PH, Liu SH, Weng CH, Lee CC, Yen TH, Chen YC, Wu TC. Risk Factors for Development of Septic Shock in Patients with Urinary Tract Infection. Biomed Res Int. 2015;2015:717094. doi: 10.1155/2015/717094. Epub 2015 Aug 25. PMID 26380292
- [Background] Simmering JE, Cavanaugh JE, Polgreen LA, Polgreen PM. Warmer weather as a risk factor for hospitalisations due to urinary tract infections. Epidemiol Infect. 2018 Feb;146(3):386-393. doi: 10.1017/S0950268817002965. Epub 2018 Jan 8. PMID 29307331
- [Background] Anderson JE. Seasonality of symptomatic bacterial urinary infections in women. J Epidemiol Community Health. 1983 Dec;37(4):286-90. doi: 10.1136/jech.37.4.286. PMID 6655418
- [Background] Kolman KB. Cystitis and Pyelonephritis: Diagnosis, Treatment, and Prevention. Prim Care. 2019 Jun;46(2):191-202. doi: 10.1016/j.pop.2019.01.001. PMID 31030820
- See also: A Diagnostics Solution Company — http://pathnostics.com